CLINICAL TRIAL: NCT02056912
Title: Identification of a New Gene Involved in Hereditary Lipodystrophy - LIPOGENE
Brief Title: Identification of a New Gene Involved in Hereditary Lipodystrophy
Acronym: LIPOGENE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CHUBX 2013/13
Record Dates: First submitted 2014-01-24; First posted 2014-02-06 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Lipodystrophy
Keywords: lipodystrophy; gene; inborn error of metabolism
MeSH Terms: conditions — Lipodystrophy; Metabolism, Inborn Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lipodystrophie Héréditaire (Other)
  Interventions: Genetic: Amplification by PCR and direct sequencing on the entire coding sequence and intron-exons boundaries of the candidate gene; Biological: Perform blood cells and fibroblasts biochemical and immuno-labeled investigations

INTERVENTIONS:
Genetic: Amplification by PCR and direct sequencing on the entire coding sequence and intron-exons boundaries of the candidate gene
Biological: Perform blood cells and fibroblasts biochemical and immuno-labeled investigations — Performed only in the two index patients enrolled in the sub-study

SUMMARY:
Human lipodystrophies (lipoD) represent a heterogeneous group of diseases characterized by generalized or partial fat loss, with fat hypertrophy in other depots when partial.3, 4 Insulin resistance, dyslipidemia and diabetes are generally associated, leading to early complications. Acquired lipoD can be generalized, resembling congenital forms, or partial, as the Barraquer-Simons syndrome, with loss of fat in the upper part of the body contrasting with accumulation in the lower part. The most common forms of lipoD are iatrogenic. In human immunodeficiency virus-infected patients, some first-generation antiretroviral drugs were strongly related with peripheral lipoatrophy and metabolic alterations. Genetic forms are very uncommon: recessive generalized congenital lipoD result in most cases from mutations in the genes encoding seipin or the 1-acyl-glycerol-3-phosphate-acyltransferase 2 (AGPAT2). Dominant partial familial lipoD result from mutations in genes encoding the nuclear protein lamin A/C or the adipose transcription factor PPARgamma. Importantly, LMNA mutations are also responsible for metabolic laminopathies, resembling the metabolic syndrome and progeria, a syndrome of premature aging. Molecular genetic bases of many rare forms of genetic lipoD remain to be elucidated.

DETAILED DESCRIPTION:
The investigators have recently evaluated two sisters (index patients) affected by a syndrome associating diffuse leukoencephalopathy and partial lipoD. The investigators have analyzed numerous known genetic causes of leukodystrophies and lipoD but the investigators failed to identify a known cause for this syndrome which has never been previously reported. The investigators then switched their effort to analyses of exome using next generation sequencing in both affected sisters and their unaffected relatives (one sister and two parents). The investigators identified an excellent candidate gene with a homozygous missense mutation in both affected sisters. The investigators now aim to prove the involvement of this candidate gene in lipoD's determinism by a search of additional mutations in the candidate gene in a series of patients affected with lipoD (collaboration with Pr Capeau's Team) (LIPOGENE study) and by functional analyses performed in the two index patients on blood and skin samples (LIPOGENE sub-study).

ELIGIBILITY:
Inclusion Criteria:

Study :

* Patients affected by lipoD
* No identified genetic cause of lipoD
* Child or adult
* DNA already available in the French reference laboratory for the genetic diagnosis of lipoD (laboratoire de Biochimie du CHU Saint-Antoine, Paris) or in the INSERM UMRS 938 laboratory, Faculté de médecine Pierre et Marie Curie Site Saint-Antoine, Paris
* Subject affiliated to the french Sécurité Sociale
* Signed consent obtained for the molecular diagnosis of lipoD.

Sub-study:

* Signed consent obtained for this sub-study from both index patients

Exclusion Criteria:

Study:

* Identified genetic cause of lipoD
* No signed consent by the patient
* Subject not affiliated to the french Sécurité Sociale.

Sub-study:

* Absence of signed consent obtained for this sub-study from both index patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Additional mutation in the studied candidate gene XX | 6 months
  Study's primary outcome
Altered lipids composition in blood red cells membranes | 6 months
  Sub-study's primary outcome
Quantitative or qualitative variation of the protein encoded by the candidate gene in fibroblasts | 6 months
  Sub-study's primary outcome
Dense deposits in fibroblasts cytoplasm | 6 months
  Sub-study's primary outcome
Phospholipids anomalies in plasma | 6 months
  Sub-study's primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure VUILLAUME, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Service de Génétique Médicale, Bordeaux, France